CLINICAL TRIAL: NCT04218721
Title: Implementing eHealth Interventions Into Regular Clinical Practice to Enhance Care Planning, Communication and Patient Involvement
Brief Title: Implementing eHealth Interventions Into Regular Clinical Practice
Acronym: InvolveMe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Nurses Organisation (Other)
Responsible Party: Principal Investigator, Elin Børøsund, Head of Research and Education, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/201
Record Dates: First submitted 2020-01-03; First posted 2020-01-06 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Renal Transplant Recipients; Non-functioning Pituitary Adenoma
Keywords: Symptom assessment; eHealth; Implementation; Communication; Shared decision making
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: All participants get access to the ehealth application
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eHealth application (Experimental): Participants get access to the eHealth application InvolveMe
  Interventions: Other: InvolveMe

INTERVENTIONS:
Other: InvolveMe — An eHealth application that allows participants to report symptoms and needs prior to out-patient visits at the hospital. The application creates a summary that allows patients to prioritize what is important to talk with their health care providers about. Health care providers can use the summary to prepare the consultation.

SUMMARY:
The purpose with this study is to test a digital patient-provider communication tool for symptom and needs management among patients with chronic health conditions.

DETAILED DESCRIPTION:
Living with chronic health conditions affects all areas of life. Fatigue, sleeping problems, pain and loneliness are common. In addition to troublesome symptoms that vary in intensity, many experience worry and uncertainty. There is a need to improve the quality of follow-up of patients with chronic health conditions. A digital patient-provider communication tool, which supports shared decision making, can be one way to improve quality.

The digital tool (InvolveMe) will provide patients with the opportunity to complete and submit a symptom and need assessment prior to out-patient visits at the hospital. Also, patients will have the opportunity to use secure e-mail for follow-up from health care providers in between hospital visits. The assessment will allow patient to prioritize what is important to talk with their health care providers about.

Such a tool can help to make changes in symptoms more visible to both patients and health care providers, as well as make it easier to ask for information and guidance to deal with the individual difficulties patients' experience. The goal is to better address symptoms and concerns and to enhance follow up and coordination between consultations as well as increase the quality of life and reduce illness related stress.

The digital communication tool is tested in a feasibility pilot study, including 23 patients with non-functioning pituitary adenomas. Participants will be given the opportunity to use the digital communication tool with baseline measures and following measures after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Non functioning pituitary adenomas (NFPA)
* Able to read and speak Norwegian
* Have access to a Smart-phone or tablet
* Have their own secure access device (BankID).

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Change in SF-36 Item Short Form Health Survey (RAND-36 version) | Baseline and 3 months
  36 item scale measuring health related quality of life (HRQoL). The scale has 8 subscales and 1 single item score. Scale and single item range: 0 to 100. Higher scores indicate higher HRQoL.
Change in The Hospital Anxiety and Depression Scale (HADS) | Baseline and 3 months
  14 item scale measuring anxiety and depression. The Scale has a total score with a scale range of 0 to 42 and an anxiety (HADS-A) and a depression (HADS-D) subscale, both with scale range of 0 to 21. Higher scores indicate higher levels of anxiety and depression

SECONDARY OUTCOMES:
Health Literacy Questionnaire (HLQ) | Baseline and 3 months
  44 item scale measuring health literacy. The scale consists of 9 subscales that covers distinct areas of health literacy. The scores for the first 5 scales range from 1 to 4, and the scores for scale 6-9 range from 1 to 5. Higher scores indicate better health literacy.

OTHER OUTCOMES:
System Usability Scale (SUS) | 3 months
  10 item scale measuring system usability. The scale has a total score with a range from 0 to 100. Higher scores indicate higher system usability.

CONTACTS AND LOCATIONS:
Overall Officials: Elin Børøsund, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seljelid B, Varsi C, Solberg Nes L, Oystese KA, Borosund E. Feasibility of a Digital Patient-Provider Communication Intervention to Support Shared Decision-Making in Chronic Health Care, InvolveMe: Pilot Study. JMIR Form Res. 2022 Apr 7;6(4):e34738. doi: 10.2196/34738. PMID 35389356
- [Background] Seljelid B, Varsi C, Solberg Nes L, Stenehjem AE, Bollerslev J, Borosund E. Content and system development of a digital patient-provider communication tool to support shared decision making in chronic health care: InvolveMe. BMC Med Inform Decis Mak. 2020 Mar 4;20(1):46. doi: 10.1186/s12911-020-1065-8. PMID 32131808
- [Background] Seljelid B, Varsi C, Solberg Nes L, Oystese KA, Borosund E. A Digital Patient-Provider Communication Intervention (InvolveMe): Qualitative Study on the Implementation Preparation Based on Identified Facilitators and Barriers. J Med Internet Res. 2021 Apr 8;23(4):e22399. doi: 10.2196/22399. PMID 33830063
- See also: Study homepage — http://involveme.no